CLINICAL TRIAL: NCT01942343
Title: Etude de l'Effet du dropéridol et de l'Ondansetron Sur l'Incidence de l'Akathisie Post opératoire en Chirurgie Ambulatoire
Brief Title: Akathisia in Post Operative Outpatients Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5505
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Akathisia
MeSH Terms: conditions — Psychomotor Agitation | interventions — Organization and Administration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 : Droperidol 1,25 mg (Active Comparator)
  Interventions: Drug: Droperidol 1,25 mg administration, Droperidol 0,625 mg administration, Odansetron 4 mg administration
- Arm 2 : Droperidol 0,625 mg (Active Comparator)
  Interventions: Drug: Droperidol 1,25 mg administration, Droperidol 0,625 mg administration, Odansetron 4 mg administration
- Arm 3 : Odansetron 4 mg (Active Comparator)
  Interventions: Drug: Droperidol 1,25 mg administration, Droperidol 0,625 mg administration, Odansetron 4 mg administration

INTERVENTIONS:
Drug: Droperidol 1,25 mg administration, Droperidol 0,625 mg administration, Odansetron 4 mg administration

SUMMARY:
The main objective of this study is to evaluate the incidence of akathisia with Droperidol, the prophylactic treatment of post operative nausea and vomiting, used at two different doses, versus control group (Ondansetron), in outpatient surgery.The primary endpoint is to compare the number of observed akathisia (Barnes score > 1) in the Droperidol arms (0,625 mg and 1,25 mg) versus Ondansetron 4 hours after recovery from anesthesia.The assumption is that there is a greater risk of akathisia among patients taking Droperidol in prevention of NPVO, that among patients taking Ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 and under 65 year-old
* Having a moderate to severe POVN (post operative vomiting and nausea) risk, meaning with at least two risk factors in the simplified Apfel score
* Outpatient surgery associated to a general anesthesia
* Patient having signed an informed consent- Patient having a social protection

Exclusion Criteria:

* Contraindication to Droperidol
* Contraindication to Ondansetron
* Patients usually treated with benzodiazepine or having been treated with benzodiazepine within 2 days prior to anesthesia
* Psychiatric and Neurodegenerative diseases
* Severe Anxiety
* Contraindication to general anesthesia or one of its components
* Allergy to propofol
* Inability to get informed (patient in an emergency situation, difficulties to understand)
* Patient under judicial protection
* Patient under tutorship or curatorship
* Pregnancy reported by the patient- Breastfeeding
* Patient in an exclusion period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of akathisia | 1 day
  The main objective of this study was to evaluate the incidence of akathisia with the waning of prophylactic treatment of PONV with droperidol used two different doses versus control group (ondansetron), ambulatory surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France

REFERENCES:
- [Result] Charton A, Greib N, Ruimy A, Faitot V, Noudem Y, Joshi GP, Meyer N, Diemunsch P. Incidence of akathisia after postoperative nausea and vomiting prophylaxis with droperidol and ondansetron in outpatient surgery: A multicentre controlled randomised trial. Eur J Anaesthesiol. 2018 Dec;35(12):966-971. doi: 10.1097/EJA.0000000000000821. PMID 29746373